CLINICAL TRIAL: NCT00509145
Title: A Multinational, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study, to Evaluate the Safety, Tolerability and Efficacy of Daily Oral Administration of Laquinimod 0.6 mg in Subjects With RRMS
Brief Title: Safety and Efficacy of Orally Administered Laquinimod Versus Placebo for Treatment of Relapsing Remitting Multiple Sclerosis (RRMS)
Acronym: ALLEGRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-LAQ-301; EUDRACT 2007-003226-19
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing; Remitting
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laquinimod (Experimental): Laquinimod 0.6 mg, oral
  Interventions: Drug: Laquinimod
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Laquinimod — Laquinimod 0.6 mg capsule, oral, once daily
  Other Names: TV-5600
  Arms: Laquinimod
Other: Placebo — oral, once daily, capsule
  Arms: Placebo

SUMMARY:
Determination the efficacy of daily oral treatment with laquinimod 0.6 mg capsules as compared to placebo in subjects with Relapsing Remitting Multiple Sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a confirmed and documented MS diagnosis as defined by the Revised McDonald criteria [Ann Neurol 2005: 58:840-846], with a relapsing-remitting disease course.
2. Subjects must be ambulatory with converted Kurtzke EDSS score of 0-5.5.
3. Subjects must be in a stable neurological condition and free of corticosteroid treatment [intravenous (iv), intramuscular (im) and/or per os (po)] 30 days prior to screening (month -1).
4. Subjects must have had experienced one of the following:

   * At least one documented relapse in the 12 months prior to screening
   * At least two documented relapses in the 24 months prior to screening
   * One documented relapse between 12 and 24 months prior to screening with at least one documented T1-Gd enhancing lesion in an MRI performed within 12 months prior to screening.
5. Subjects must be between 18 and 55 years of age, inclusive.
6. Subjects must have disease duration of at least 6 months (from the first symptom) prior to screening.
7. Women of child-bearing potential must practice an acceptable method of birth control [acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy or double-barrier method (condom or diaphragm with spermicide).
8. Subjects must be able to sign and date a written informed consent prior to entering the study
9. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

1. Subjects with progressive forms of MS
2. An onset of relapse, unstable neurological condition or any treatment with corticosteroids [intravenous (iv), intramuscular (im) and/or per os (po)] or ACTH between month -1 (screening) and 0 (baseline).
3. Use of experimental or investigational drugs, and/or participation in drug clinical studies within the 6 months prior to screening.
4. Use of immunosuppressive including Mitoxantrone (Novantrone®) or cytotoxic agents within 6 months prior to the screening visit.
5. Previous use of either of the following: natalizumab (Tysabri®), cladribine, laquinimod.
6. Previous treatment with glatiramer acetate (Copaxone®) Interferon-β (either 1a or 1b) or IVIG within 2 months prior to screening visit.
7. Systemic corticosteroid treatment of ≥30 consecutive days duration within 2 months prior to screening visit.
8. Previous total body irradiation or total lymphoid irradiation.
9. Previous stem cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
10. A known history of tuberculosis.
11. Acute infection two weeks prior to baseline visit.
12. Major trauma or surgery two weeks prior to baseline
13. A history of vascular thrombosis (excluding catheter-site superficial venous thrombophlebitis).
14. A carrier state of factor V Leiden mutation (either homo- or heterozygous) as disclosed at screening.
15. Positive screening test for Hepatitis B surface antigen, Hepatitis C antibody, or HIV antibody as disclosed at screening visit.
16. Use of potent inhibitors of CYP3A4 within 2 weeks prior to baseline visit (1 month for fluoxetine) see detailed list in Appendix 5
17. Use of amiodarone within 2 years prior to screening visit.
18. Pregnancy or breastfeeding.
19. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical examinations, ECG, laboratory tests or chest X-ray. Such conditions may include:

    * A cardiovascular or pulmonary disorder that cannot be well-controlled by standard treatment permitted by the study protocol.
    * A gastrointestinal disorder that may affect the absorption of study medication.
    * Renal or metabolic diseases.
    * Any form of chronic liver disease, including known non-alcoholic steatohepatitis.
    * A ≥2xULN serum elevation of either of the following at screening: ALT, AST or direct bilirubin
    * A QTC interval (obtained from either 2 ECG recordings at screening or from the mean value calculated from 3 measurements at baseline visit) which is >450msec.
    * A family history of Long- QT syndrome.
    * A history of drug and/or alcohol abuse.
    * Major psychiatric disorder.
20. A known history of sensitivity to Gd.
21. Inability to successfully undergo MRI scanning.
22. Known drug hypersensitivity that would preclude administration of laquinimod, such as hypersensitivity to: mannitol, meglumine or sodium stearyl fumarate.

Exclusion Criteria:

1. Subjects who suffer from any form of progressive MS.
2. Any condition which the investigator feels may interfere with participation in the study.
3. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation,
4. Subjects who received any investigational medication, immunosuppressives or cytotoxic agents within 6 months prior to screening
5. Previous treatment with immunomodulators within two months prior to screening
6. Pregnancy or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1106 (Actual)
Dates: Start 2007-11-13 (Actual); Primary Completion 2010-11-08 (Actual); Study Completion 2010-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, Principal Investigator — U.O.Neurology-Neurorehabilitation and Clinical Neurophysiology
Locations (144):
- United States (23):
  - Teva Investigational Site 1076, Phoenix, Arizona
  - Teva Investigational Site 1090, Centennial, Colorado
  - Teva Investigational Site 1088, Fort Collins, Colorado
  - Teva Investigational Site 1094, New Haven, Connecticut
  - Teva Investigational Site 1102, Northbrook, Illinois
  - Teva Investigational Site 1081, Fort Wayne, Indiana
  - Teva Investigational Site 1083, Des Moines, Iowa
  - Teva Investigational Site 1086, Kansas City, Kansas
  - Teva Investigational Site 1101, Lexington, Kentucky
  - Teva Investigational Site 1096, Farmington Hills, Michigan
  - Teva Investigational Site 1093, Minneapolis, Minnesota
  - Teva Investigational Site 1098, St Louis, Missouri
  - Teva Investigational Site 1082, New York, New York
  - Teva Investigational Site 1079, Rochester, New York
  - Teva Investigational Site 1073, Winston-Salem, North Carolina
  - Teva Investigational Site 1097, Fargo, North Dakota
  - Teva Investigational Site 1084, Dayton, Ohio
  - Teva Investigational Site 1092, Oklahoma City, Oklahoma
  - Teva Investigational Site 1100, Hershey, Pennsylvania
  - Teva Investigational Site 1087, Philadelphia, Pennsylvania
  - Teva Investigational Site 1075, Lubbock, Texas
  - Teva Investigational Site 1078, San Antonio, Texas
  - Teva Investigational Site 1085, Milwaukee, Wisconsin
- Austria (4):
  - Teva Investigational Site 3300, Klagenfurt
  - Teva Investigational Site 3303, Linz
  - Teva Investigational Site 3302, Sankt Pölten
  - Teva Investigational Site 3301, Villach
- Bulgaria (6):
  - Teva Investigational Site 5901, Pleven
  - Teva Investigational Site 5904, Sofia
  - Teva Investigational Site 5903, Sofia
  - Teva Investigational Site 5900, Sofia
  - Teva Investigational Site 5905, Sofia
  - Teva Investigational Site 5902, Varna
- Canada (7):
  - Teva Investigational Site 1132, Halifax, Nova Scotia
  - Teva Investigational Site 1126, London, Ontario
  - Teva Investigational Site 1128, Ottawa, Ontario
  - Teva Investigational Site 1134, Toronto, Ontario
  - Teva Investigational Site 1130, Greenfield Park, Quebec
  - Teva Investigational Site 1129, Montreal, Quebec
  - Teva Investigational Site 1131, Sherbrooke, Quebec
- Czechia (2):
  - Teva Investigational Site 5417, Olomouc
  - Teva Investigational Site 5416, Ostrava - Poruba
- Estonia (2):
  - Teva Investigational Site 5504, Tallinn
  - Teva Investigational Site 5505, Tartu
- France (6):
  - Teva Investigational Site 3525, Besançon
  - Teva Investigational Site 3527, Bron
  - Teva Investigational Site 3526, Clermont-Ferrand
  - Teva Investigational Site 3524, Lille
  - Teva Investigational Site 3528, Marseille
  - Teva Investigational Site 3529, Rennes
- Georgia (2):
  - Teva Investigational Site 8100, Tbilisi
  - Teva Investigational Site 8101, Tbilisi
- Germany (16):
  - Teva Investigational Site 3247, Bayreuth
  - Teva Investigational Site 3241, Berlin
  - Teva Investigational Site 3238, Berlin
  - Teva Investigational Site 3248, Bochum
  - Teva Investigational Site 3245, Dresden
  - Teva Investigational Site 3237, Emden
  - Teva Investigational Site 3242, Erbach im Odenwald
  - Teva Investigational Site 3240, Erfurt
  - Teva Investigational Site 3249, Freiburg im Breisgau
  - Teva Investigational Site 3236, Hamburg
  - Teva Investigational Site 3246, Hamburg
  - Teva Investigational Site 3239, Hanover
  - Teva Investigational Site 3243, Heidelberg
  - Teva Investigational Site 3251, Münster
  - Teva Investigational Site 3250, Trier
  - Teva Investigational Site 3244, Ulm
- Hungary (4):
  - Teva Investigational Site 5115, Budapest
  - Teva Investigational Site 5114, Debrecen
  - Teva Investigational Site 5116, Miskolc
  - Teva Investigational Site 5117, Veszprém
- Israel (5):
  - Teva Investigational Site 8034, Haifa
  - Teva Investigational Site 8031, Haifa
  - Teva Investigational Site 8030, Jerusalem
  - Teva Investigational Site 8033, Ramat Gan
  - Teva Investigational Site 8032, Tel Aviv
- Italy (10):
  - Teva Investigational Site 3044, Catania
  - Teva Investigational Site 3045, Fidenza
  - Teva Investigational Site 3042, Gallarate
  - Teva Investigational Site 3046, Grosseto
  - Teva Investigational Site 3047, Milan
  - Teva Investigational Site 3038, Milan
  - Teva Investigational Site 555, Milan
  - Teva Investigational Site 3039, Milan
  - Teva Investigational Site 3041, Palermo
  - Teva Investigational Site 3040, Rome
- Teva Investigational Site 5604, Riga, Latvia
- Lithuania (2):
  - Teva Investigational Site 5704, Kaunas
  - Teva Investigational Site 5705, Šiauliai
- Netherlands (3):
  - Teva Investigational Site 3809, Groesbeek
  - Teva Investigational Site 3810, Nieuwegein
  - Teva Investigational Site 3811, Tilburg
- Poland (8):
  - Teva Investigational Site 5322, Częstochowa
  - Teva Investigational Site 5319, Gmina Końskie
  - Teva Investigational Site 5320, Gorzów Wielkopolski
  - Teva Investigational Site 5316, Katowice
  - Teva Investigational Site 5318, Kielce
  - Teva Investigational Site 5317, Krakow
  - Teva Investigational Site 5315, Lodz
  - Teva Investigational Site 5325, Warsaw
- Romania (5):
  - Teva Investigational Site 5208, Bucharest
  - Teva Investigational Site 5210, Cluj-Napoca
  - Teva Investigational Site 5212, Constanța
  - Teva Investigational Site 5211, Târgu Mureş
  - Teva Investigational Site 5209, Timișoara
- Russia (11):
  - Teva Investigational Site 5031, Kemerovo
  - Teva Investigational Site 5021, Moscow
  - Teva Investigational Site 5028, Nizhny Novgorod
  - Teva Investigational Site 5027, Novosibirsk
  - Teva Investigational Site 5030, Perm
  - Teva Investigational Site 5026, Saint Petersburg
  - Teva Investigational Site 5025, Saint Petersburg
  - Teva Investigational Site 5024, Saint Petersburg
  - Teva Investigational Site 5022, Saint Petersburg
  - Teva Investigational Site 5023, Saint Petersburg
  - Teva Investigational Site 5029, Yekaterinburg
- Serbia (2):
  - Teva Investigational Site 6100, Belgrade
  - Teva Investigational Site 6102, Niš
- Spain (13):
  - Teva Investigational Site 3132, Barcelona
  - Teva Investigational Site 3134, Barcelona
  - Teva Investigational Site 3144, Barcelona
  - Teva Investigational Site 3140, Beade-Vigo
  - Teva Investigational Site 3142, Getafe
  - Teva Investigational Site 3136, Girona
  - Teva Investigational Site 3135, Lleida
  - Teva Investigational Site 3133, Madrid
  - Teva Investigational Site 3146, Madrid
  - Teva Investigational Site 3137, Murcia
  - Teva Investigational Site 3138, Pontevedra
  - Teva Investigational Site 3139, Santiago de Compostela
  - Teva Investigational Site 3143, Valencia
- Sweden (3):
  - Teva Investigational Site 4204, Stockholm
  - Teva Investigational Site 4205, Stockholm
  - Teva Investigational Site 4206, Stockholm
- Teva Investigational Site 8201, Izmir, Turkey (Türkiye)
- Ukraine (5):
  - Teva Investigational Site 5803, Dnipropetrovsk
  - Teva Investigational Site 5802, Kyiv
  - Teva Investigational Site 5804, Kyiv
  - Teva Investigational Site 5800, Lviv
  - Teva Investigational Site 5801, Vinnytsia
- United Kingdom (3):
  - Teva Investigational Site 3425, Liverpool
  - Teva Investigational Site 3424, London
  - Teva Investigational Site 3422, Sheffield

REFERENCES:
- [Derived] Kolb-Sobieraj C, Gupta S, Weinstock-Guttman B. Laquinimod therapy in multiple sclerosis: a comprehensive review. Neurol Ther. 2014 May 6;3(1):29-39. doi: 10.1007/s40120-014-0017-6. eCollection 2014 Jun. PMID 26000222
- [Derived] Filippi M, Rocca MA, Pagani E, De Stefano N, Jeffery D, Kappos L, Montalban X, Boyko AN, Comi G; ALLEGRO Study Group. Placebo-controlled trial of oral laquinimod in multiple sclerosis: MRI evidence of an effect on brain tissue damage. J Neurol Neurosurg Psychiatry. 2014 Aug;85(8):851-8. doi: 10.1136/jnnp-2013-306132. Epub 2013 Sep 12. PMID 24029546
- [Derived] Comi G, Jeffery D, Kappos L, Montalban X, Boyko A, Rocca MA, Filippi M; ALLEGRO Study Group. Placebo-controlled trial of oral laquinimod for multiple sclerosis. N Engl J Med. 2012 Mar 15;366(11):1000-9. doi: 10.1056/NEJMoa1104318. PMID 22417253
- See also: Teva's Allegro Clinical Trials website — http://www.TevaClinicalTrials.com/patients/default.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1106 participants were enrolled and randomized in the placebo-controlled (PC) double-blind period. Participants were randomized 1:1 to the treatment arms.
Groups:
- Laquinimod: Laquinimod 0.6 mg capsule taken orally once a day
- Placebo: Matching placebo capsule taken orally once a day
Period: Overall Study
Arm/Group | Laquinimod | Placebo
Started | 550 | 556
Completed | 437 | 427
Not Completed | 113 | 129
Not completed — Death | 0 | 2
Not completed — Adverse Event | 42 | 28
Not completed — Withdrawal by Subject | 32 | 38
Not completed — Physician Decision | 11 | 14
Not completed — Protocol Violation | 1 | 6
Not completed — Pregnancy | 3 | 8
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by participant after confirmed relapse | 12 | 22
Not completed — Other | 6 | 6

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all participants that were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Laquinimod | Placebo | Total
Number analyzed (Participants) | 550 | 556 | 1106
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (9.2) | 38.5 (9.1) | 38.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 391 | 368 | 759
  Male | 159 | 188 | 347
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Race not reported for 4 participants.
  Participants
    Race : Asian: number analyzed (Participants) | 548 | 554 | 1102
    Race : Asian | 2 | 1 | 3
    Race : Black or African American: number analyzed (Participants) | 548 | 554 | 1102
    Race : Black or African American | 1 | 8 | 9
    Race : White: number analyzed (Participants) | 548 | 554 | 1102
    Race : White | 532 | 532 | 1064
    Race : Hispanic: number analyzed (Participants) | 548 | 554 | 1102
    Race : Hispanic | 11 | 9 | 20
    Race : Other: number analyzed (Participants) | 548 | 554 | 1102
    Race : Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Relapse Rate: Number of Confirmed Relapses During the Double Blind Study Period
Description: A relapse was defined as the appearance of at least one new neurological abnormality or the reappearance of at least one previously observed neurological abnormalities lasting greater than or equal to 48 hours and immediately preceded by an improving neurological state of greater than or equal to 30 days from onset of previous relapse. An event was counted as a relapse only when the participant's symptoms were accompanied by observed objective neurological changes, consistent with one or more of the following: An increase of greater than or equal to 0.5 in the Expanded Disability Status Scale (EDSS) score as compared to previous evaluation, an increase of one grade in the actual score of greater than or equal to 2 of the 7 functional systems (FS), as compared to previous evaluation, or an increase of 2 grades in the actual score of one FS as compared to the previous evaluation.
Time Frame: Up to Month 24
Population: Intent to treat (ITT) analysis set included all randomized participants.
Measure: Mean (Standard Deviation); unit: Confirmed relapses
Arm/Group | Laquinimod | Placebo
Number analyzed (Participants) | 550 | 556
Confirmed relapses | 0.54 (0.88) | 0.67 (0.92)
Statistical Analysis 1: Comparison: Laquinimod vs Placebo; Response variable: number of relapses during 24 months. Offset based on the log of subject's exposure in years was employed to adjust for variability of treatment exposure. In addition to the treatment group, the Poisson regression model included the following covariates: baseline EDSS score, log of prior 2-year number of relapses+1 and Country or Geographical Region (CGR); Test type: Superiority; p = 0.0024, Over-dispersed Poisson Regression; Risk Ratio (RR) = 0.770, 95% CI 2-sided [0.650 to 0.911], Standard Error of Mean 0.066 — Laquinimod 0.6 mg vs. placebo

2. Secondary Outcome: Composite Endpoint: Sum of the Number of T1 Gadolinium (Gd)-Enhanced Lesions on T1-Weighted MRI Images
Description: Composite score was calculated as the sum of the number of gadolinium (Gd)-enhanced lesions at Month 12 and the number of gadolinium (Gd)-enhanced lesions at Month 24 on T1-Weighted MRI scans.
Time Frame: Month 12, Month 24
Population: ITT analysis set included all randomized participants. Number of participants analyzed included the number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Laquinimod | Placebo
Number analyzed (Participants) | 482 | 464
Lesions | 1.86 (5.02) | 2.92 (7.58)

3. Secondary Outcome: Composite Endpoint: Sum of the Number of New/Enlarging T2 Lesions
Description: Composite score calculated as the sum of T2 lesions at Months 12 and 24 that are new or enlarged.
Time Frame: Month 12, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Laquinimod | Placebo
Number analyzed (Participants) | 482 | 464
Lesions | 5.26 (9.08) | 7.87 (12.56)

4. Secondary Outcome: Accumulation of Physical Disability Measured by the Time to Confirmed Progression of Expanded Disability Status Scale (EDSS)
Description: EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]). A confirmed progression of EDSS is defined as at least 1 point increase from baseline if baseline EDSS was between 0 and 5.0, or at least 0.5 point increase if baseline EDSS was 5.5 or higher, confirmed 3 months later. Participants were assessed between baseline and month 24 visit. Participants that met these criteria for any 3 consecutive months were counted in the progression category. Progression could not be confirmed during an MS relapse. Data is presented as a distribution of confirmed disease progression (CDP) events (number of participants with CDP).
Time Frame: Baseline to Month 24
Population: ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Laquinimod | Placebo
Number analyzed (Participants) | 550 | 556
Participants
  Progressed | 54 | 78
  Progression Free | 496 | 478

5. Secondary Outcome: Change From Baseline in Disability as Assessed by the Multiple Sclerosis Functional Composite (MSFC) Score
Description: The Multiple Sclerosis Functional Composite is an instrument assessing disability that consists of 3 clinical assessments. The 3 are Timed 25-Foot Walk, 9-Hole Peg Test which measures upper extremity (arm and hand) function, and PASAT (Paced Auditory Serial Addition Test) which is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. A Z-score is used to define a common metric from the 3 assessments that constitute the MSFC score. The study's population at baseline was used as reference population for the Z-score calculation. A Z-score of 0 represents the population mean at baseline. Higher Z-scores correspond to an improved outcome.
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Laquinimod | Placebo
Number analyzed (Participants) | 424 | 420
Z score | 0.0 (0.4) | 0.0 (0.7)

ADVERSE EVENTS:
Time Frame: Baseline to 24 months
Description: Safety analysis included all participants that received at least one dose of study drug.
Groups:
- Laquinimod 0.6 mg: Laquinimod 0.6 mg capsule taken orally once a day
Arm/Group | Laquinimod 0.6 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/550 | 3/556
Serious Adverse Events (participants affected / at risk) | 61/550 | 53/556
Other Adverse Events (participants affected / at risk) | 368/550 | 346/556
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laquinimod 0.6 mg (N=550) | Placebo (N=556)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (4) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (4)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 5 (5) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 2 (2) | 5 (7)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Hysterectomy (Surgical and medical procedures) | 2 (2) | 4 (4)
Spinal fusion surgery (Surgical and medical procedures) | 2 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug interaction (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (2) | 0 (0)
Staphylococcal pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Bacterial test positive (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian granulosa-theca cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Fallopian tube cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian adhesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine cervical squamous metaplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 1 (1)
Anorectal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Bone graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Bone operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholesteatoma removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Chondroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Cyst drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Ligament operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Plasmapheresis (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 3 (3)
Renal stone removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Turbinectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Uterine dilation and curettage (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Vein disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laquinimod 0.6 mg (N=550) | Placebo (N=556)
Abdominal pain upper (Gastrointestinal disorders) | 28 (33) | 29 (34)
Diarrhoea (Gastrointestinal disorders) | 42 (49) | 33 (41)
Nausea (Gastrointestinal disorders) | 34 (38) | 32 (38)
Fatigue (General disorders) | 25 (28) | 29 (36)
Influenza (Infections and infestations) | 33 (39) | 44 (50)
Nasopharyngitis (Infections and infestations) | 100 (159) | 119 (199)
Sinusitis (Infections and infestations) | 29 (40) | 25 (38)
Upper respiratory tract infection (Infections and infestations) | 42 (61) | 48 (62)
Urinary tract infection (Infections and infestations) | 40 (60) | 24 (35)
Alanine aminotransferase increased (Investigations) | 38 (49) | 15 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 (61) | 41 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 89 (122) | 50 (73)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 35 (47) | 38 (44)
Headache (Nervous system disorders) | 123 (225) | 99 (176)
Depression (Psychiatric disorders) | 30 (31) | 32 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (47) | 25 (29)
Abdominal pain (Gastrointestinal disorders) | 31 (36) | 15 (16)
Pyrexia (General disorders) | 20 (21) | 28 (34)
Dizziness (Nervous system disorders) | 27 (29) | 29 (33)
Insomnia (Psychiatric disorders) | 36 (40) | 31 (39)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 (24) | 29 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.